CLINICAL TRIAL: NCT06638502
Title: Double Blind, Randomized, Placebo Controlled, Study to Evaluate the Safety of HRX215 in Patients Post Major Hepatectomy, Preceded by an Open Pilot Phase in Patients Post Minor Hepatectomy Due to Metastases of a Colon Carcinoma
Brief Title: Safety of HRX215 in Patients After Minor and Major Liver Resection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HepaRegeniX GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRX215-CR03-LR01
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Liver Metastases; Liver Resection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active treatment minor hepatic resection (Experimental): 5 participants will receive HRX215 250 mg twice daily orally within 1-3 days after minor (<=31%) liver resection for colorectal liver metastases for 28 days.
  Interventions: Drug: HRX215 capsules
- Active treatment arm major hepatic resection (Active Comparator): 10 participants will receive HRX215 250 mg twice daily orally within 1-3 days after major (50-72%) liver resection for colorectal liver metastases for 28 days.
  Interventions: Drug: HRX215 capsules
- placebo arm major hepatic resection (Placebo Comparator): 10 participants will receive placebo capsules with matching appearance to HRX215 twice daily orally within 1-3 days after major (50-72%) liver resection for colorectal liver metastases for 28 days
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: HRX215 capsules — HRX215 capsules 250 mg orally twice daily
  Arms: Active treatment arm major hepatic resection; Active treatment minor hepatic resection
Drug: Placebo capsules — placebo capsules matching appearance of HRX215
  Arms: placebo arm major hepatic resection

SUMMARY:
The goal of this clinical trial is to learn if HRX215 is safe and tolerable in adults who have undergone surgical removal of metastatic tumor(s) due to colorectal carcinoma in the liver.

The main question it aims to answer are:

1. to learn about the safety of HRX215
2. to learn about how the body absorbs, distributes, and gets rid of HRX215 . Researchers will compare HRX215 to a placebo (a look-alike substance that contains no drug) to see what medical problems participants have when taking HRX215.

Participants will:

Take HRX215 or a placebo twice a day for 28 days Daily visits for 7 days for checkups and tests which may either be in the hospital or outpatient after 3 days. Clinic visits every two weeks for the next two visits. The visit at two weeks may be a home visit or clinic visit. Additional clinic visits 3 months and 6 months after the start of treatment

DETAILED DESCRIPTION:
The study is designed to evaluate primarily the safety of HRX215, first after minor liver resection and, when safety is established, in those patients after major liver resection. Participants will start treatment within 1-3 days after liver resection and will receive 28 day treatment with HRX215 twice daily or placebo with follow up visits 3 and 6 months after completion of treatment.

The pharmacokinetics will be compared with the results of the phase I studies, whereas efficacy will be evaluated only descriptively. Secondary objectives will include evaluation of differences in liver volume recovery postoperatively and clinical outcomes including days in the ICU and 90 day mortality in participants who receive treatment with HRX215 vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Stable male and female patients between 18 and 75 years within 1-3 days after extended resection of the right or left liver lobe due to metastases of a colon carcinoma, but otherwise normal liver parenchyma proven by histopathology assessment of a liver biopsy within 3 months before surgery and liver functional parameters.
2. For the pilot phase less extended resections (remnant liver volume >69%) are required)
3. Percentage of Remnant Liver Volume (RLV) 28%-50% (randomized part of the study)

   -

Exclusion Criteria:

1. Liver Cirrhosis
2. Preoperative presence of clinical ascites
3. Any other liver cancer
4. BMI >35 kg/m2
5. ASA Score>4
6. CC Score >0: all patients with pre-operatively or intra-operatively diagnosed peritoneal carcinosis or other pre-op or intra-op findings which would deem the patient to be unresectable, are excluded.
7. Incomplete liver metastasis resection -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
• Adverse Events (AEs) observed. | 28 days
  * Adverse Events (AEs) observed
  * Clinical laboratory investigation including hematology, blood glucose, HbA1c, serum chemistry: pre-treatment, after 14 and 28 days

SECONDARY OUTCOMES:
Pharmacokinetic Plasma Analysis | 28 days
  Levels of drug (HRX215) at selected time intervals after drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Linda E Greenbaum, M.D., Study Director — HepaRegeniX GmbH; Patrick Starlinger, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States